CLINICAL TRIAL: NCT02254447
Title: An Open-label, Randomized, Single Dose, Three-way Crossover, Six Sequence Pilot Study to Determine the Relative Bioavailability of Candesartan Cilexetil 16mg From Two Candidate Tablet Formulations of GW615775 Relative to One 16mg Tablet of Reference Candesartan Cilexetil in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Relative Bioavailability Study of Candesartan Cilexetil Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201713
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Disease
Keywords: relative bio-availability; fasting; GW615775; Candesartan cilexetil; ATACAND
MeSH Terms: conditions — Cardiovascular Diseases; Fasting | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence ABC (Experimental): Subjects in this arm will receive single dose of treatment A in period 1, treatment B in period 2 and treatment C in period 3 (one treatment per period), where treatment A= ATACAND as a reference treatment containing Candesartan cilexetil 16 mg, treatment B= Test formulation 1 containing Candesartan cilexetil 16 mg, and treatment C= Test formulation 2 containing Candesartan cilexetil 16 mg.
  Interventions: Drug: Candesartan Cilexetil in formulation 1; Drug: Candesartan Cilexetil in formulation 2; Drug: ATACAND
- Sequence ACB (Experimental): Subjects in this arm will receive single dose of treatment A in period 1, treatment C in period 2 and treatment B in period 3 (one treatment per period), where treatment A= ATACAND as a reference treatment containing Candesartan cilexetil 16 mg, treatment B= Test formulation 1 containing Candesartan cilexetil 16 mg, and treatment C= Test formulation 2 containing Candesartan cilexetil 16 mg.
  Interventions: Drug: Candesartan Cilexetil in formulation 1; Drug: Candesartan Cilexetil in formulation 2; Drug: ATACAND
- Sequence BAC (Experimental): Subjects in this arm will receive single dose of treatment B in period 1, treatment A in period 2 and treatment C in period 3 (one treatment per period), where treatment A= ATACAND as a reference treatment containing Candesartan cilexetil 16 mg, treatment B= Test formulation 1 containing Candesartan cilexetil 16 mg, and treatment C= Test formulation 2 containing Candesartan cilexetil 16 mg.
  Interventions: Drug: Candesartan Cilexetil in formulation 1; Drug: Candesartan Cilexetil in formulation 2; Drug: ATACAND
- Sequence BCA (Experimental): Subjects in this arm will receive single dose of treatment B in period 1, treatment C in period 2 and treatment A in period 3 (one treatment per period), where treatment A= ATACAND as a reference treatment containing Candesartan cilexetil 16 mg, treatment B= Test formulation 1 containing Candesartan cilexetil 16 mg, and treatment C= Test formulation 2 containing Candesartan cilexetil 16 mg.
  Interventions: Drug: Candesartan Cilexetil in formulation 1; Drug: Candesartan Cilexetil in formulation 2; Drug: ATACAND
- Sequence CAB (Experimental): Subjects in this arm will receive single dose of treatment C in period 1, treatment A in period 2 and treatment B in period 3 (one treatment per period), where treatment A= ATACAND as a reference treatment containing Candesartan cilexetil 16 mg, treatment B= Test formulation 1 containing Candesartan cilexetil 16 mg, and treatment C= Test formulation 2 containing Candesartan cilexetil 16 mg.
  Interventions: Drug: Candesartan Cilexetil in formulation 1; Drug: Candesartan Cilexetil in formulation 2; Drug: ATACAND
- Sequence CBA (Experimental): Subjects in this arm will receive single dose of treatment C in period 1, treatment B in period 2 and treatment A in period 3 (one treatment per period), where treatment A= ATACAND as a reference treatment containing Candesartan cilexetil 16 mg, treatment B= Test formulation 1 containing Candesartan cilexetil 16 mg, and treatment C= Test formulation 2 containing Candesartan cilexetil 16 mg.
  Interventions: Drug: Candesartan Cilexetil in formulation 1; Drug: Candesartan Cilexetil in formulation 2; Drug: ATACAND

INTERVENTIONS:
Drug: Candesartan Cilexetil in formulation 1 — Round, biconvex white tablets containing Candesartan cilexetil 16 mg for oral administration
Drug: Candesartan Cilexetil in formulation 2 — Round, biconvex white tablets containing Candesartan cilexetil 16 mg for oral administration
Drug: ATACAND — Round, biconvex pink tablets containing Candesartan cilexetil 16 mg for oral administration

SUMMARY:
This study will investigate the relative bioavailability of two candidate tablet formulations of 16 milligram (mg) Candesartan cilexetil (GW615775) compared with the reference product ATACAND™ containing 16 mg Candesartan cilexetil in healthy human subjects. This is an open-label, randomized, single dose, three-way crossover, six sequence study enrolling 18 healthy human subjects to ensure at least 14 subjects complete the study as planned. Each subject enrolled will participate in all three treatment periods and will be assigned to one of the six treatment sequences, in accordance with the randomization schedule. The treatment periods will be separated by a washout period of at least 7 days and no more than 14 days between dosing occasions. A follow up visit will be conducted 14-21 days post last dosing. ATACAND is a registered trademark of the AstraZeneca group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilograms (kg) and Body Mass Index within the range 19 -24.9 kg/meter (m)^2 (inclusive).
* Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as: Pre-menopausal females with documented tubal ligation, or documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, or hysterectomy, or documented bilateral oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until [at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer] after the last dose of study medication and completion of the follow-up visit.

GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP. This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penilevaginal intercourse on a long term and persistent basis:

Contraceptive subdermal implant that meets the effectiveness criteria including a <1% rate of failure per year, as stated in the product label.

Intrauterine device or intrauterine system that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label.

Oral Contraceptive, either combined or progestogen alone. Injectable progestogen Contraceptive vaginal ring Percutaneous contraceptive patches Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository) only for the following 3 situations when there is a very low risk for developmental toxicity: Vaccines, Monoclonal antibodies when there is no target biology concern, Compounds that have a complete reproductive toxicology package and, have not shown any signal for developmental toxicity.

The investigator is responsible for ensuring that subjects understand how to properly use the following methods of contraception. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until [at least five half-lives of study medication OR for a cycle of spermatogenesis following five terminal half-lives] after the last dose of study medication: vasectomy with documentation of azoospermia, male condom plus partner use of one of the contraceptive options below:

Contraceptive subdermal implant that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label.

Oral Contraceptive, either combined or progestogen alone Injectable progestogen Contraceptive vaginal ring Percutaneous contraceptive patches

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Alanine aminotransferase and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected (QTc) > 450 millisecond (msec).
* No concomitant medications should be taken by the subject while participating in the study.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8grams of alcohol: a half-pint (equivalent to 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Hypersensitivity to candesartan cilexetil or to any of the excipients.
* Presence of hepatitis B surface antigen positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* The subject has participated in a clinical trial and has received an investigational current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* Any symptoms with a systolic blood pressure<95millimeter of mercury.
* Pregnant females as determined by positive serum human chorionic gonadotrophin test at screening or prior to dosing.
* Lactating females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters. | PK samples will be collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24, 36 and 48 hours post dose in each treatment period.
  Pharmacokinetic parameters will be measured to estimate the relative bio-availability following administration of two candidate tablet formulations of Candesartan cilexetil relative to reference Candesartan cilexetil tablet. Pharmacokinetic parameters include: maximum observed concentration (Cmax), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinite]), Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC[0-t]).

SECONDARY OUTCOMES:
Plasma PK profile | PK samples will be collected at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24, 36 and 48 hours post dose in each treatment period.
  Pharmacokinetic parameters to be estimated include: time of occurrence of Cmax (Tmax), terminal phase half-life (t1/2) and percentage of AUC(0-infinity) obtained by extrapolation (%AUCex).
Vital sign assessment as a safety measure | Up to 30 days
  Vital sign assessment include: blood pressure and pulse rate measurements.
Number of subjects with adverse events as a safety measure | 50 days
  Adverse events will be collected from the start of Study Treatment until the subject's final discharge from study at the end of Treatment Period 3, follow-up call or last outpatient visit, whichever is the latest.
Laboratory parameter assessment as a safety measure | Up to 30 days
  Laboratory parameters include: hematology, clinical chemistry, urinalysis and additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 201713 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201713?search=study&search_terms=201713#rs
- Available data/document: Individual Participant Data Set: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201713 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register